CLINICAL TRIAL: NCT07256431
Title: Environmental Risk Factors in Multiple Sclerosis Development: Epidemiological Study of EBV Infection and Vitamin D Deficiency in RIS Patients
Acronym: RIS - EBVD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2025/PROBIORIS/EBVD
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Radiologically Isolated Syndrome; Epstein-Barr Virus Infections
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma samples already in biobanks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with radiologically isolated syndrome
  Interventions: Other: Antibiody titration
- Healthy controls
  Interventions: Other: Antibiody titration

INTERVENTIONS:
Other: Antibiody titration — Search for EBV seropositivity using SIMAO assay

SUMMARY:
This is an ancillary study using samples collected in the ProBioRIS cohort (NCT06395662). The aim of the project is to highlight new biomarker candidates to assess the risk of conversion to clinically definite multiple sclerosis (CDMS) and disease activity (Evidence of Disease Activity) by taking into account demographic, clinical and MRI parameters. A cohort of healthy subjects will be integrated into the study to serve as a control population. We will study a panel of serum immunoglobulins targeting different Epstein Barr virus antigens to identify latency or reactivation phases. Identifying and prioritizing risk factors for clinical conversion to MS in radiologically isolated syndrome patients is of major importance for the implementation of personalized monitoring and treatment strategies, especially following the recent highlighting of the benefit of background treatments in patients at high risk of CDMS.

ELIGIBILITY:
Inclusion Criteria:

* RIS patients from the ProBioRIS study with sufficient serum residuals for vitamin D testing and complete EBV serology.
* Healthy subjects who participated in the VDSS trial and who provided consent for the use, for basic research purposes, of human biological samples collected during the trial.

Exclusion Criteria:

• Insufficient sample

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with RIS taken from ProBioRIS cohort (NCT06395662) plus healthy controls taken from the VDSS study (NCT05654818).
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of EBV seropositivity in RIS patients | Baseline
  Measured by single-molecule array (SIMOA)
Serum vitamin D levels in patients with RIS | Baseline
  Measured with mass spectrometry
Disease activity in patients with RIS | Baseline
  Evidence of disease aftivity versus no evidence of disease activity

SECONDARY OUTCOMES:
Prevalence of EBV seropositivity in healthy controls | Baseline
  Measured by single-molecule array (SIMOA)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvenot, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France